CLINICAL TRIAL: NCT00425724
Title: HSP-glomerulonephritis Trial: MP vs CyA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Responsible Party: Dr. Matti Nuutinen, Oulu Univ. Hospital, Oulu Univ. Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25600
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Purpura, Schoenlein-Henoch
Keywords: proteinuria; nephritis; nephrotic syndrome; glomerulonephritis
MeSH Terms: conditions — IgA Vasculitis; Proteinuria; Nephritis; Nephrotic Syndrome; Glomerulonephritis

INTERVENTIONS:
Drug: Methylprednisolone pulses plus prednisone versus Cyclosporine A — The patients will be randomised to receive either MP pulses i.v. or cyclosporine A p.o. The MP pulses will consist of three doses of methylprednisolone 30 mg/kg i.v. given over a period of one week in hospital. On the intermediate days and for a month after the MP pulses, the patients will be given prednisone 30 mg/m2/day p.o., after which the prednisone medication will be gradually run down over 3 months. The patients randomised into the cyclosporine A group will receive an initial dose of 5 mg/kg/day, after which the dosage will be titrated to an optimal therapeutic level by monitoring the B-Cya concentration. The cyclosporine A treatment will be continued for 12 months.

SUMMARY:
No curative treatment of severe HSP nephritis is known.

Apart from corticosteroids, immunosuppressive drugs, such as azathioprine and cyclophosphamide, have been used to treat severe HSP nephritis.Limited patient series treated with these drugs have been described, but there are no reports of controlled trials.

Cyclosporine A have been used to treat corticosteroid-resistant or corticosteroid-dependent nephrosis. (11) Cyclosporine A has also been used to treat HSP nephritis, but as far as we know, there are no publications reporting such trials.

The aim of the study is to compare MP pulses and cyclosporine A for their efficacy in the treatment of HSP nephritis.

The efficacy of the two treatments will be assessed on the basis of the duration of nephrosis/nephritis, the maintenance of renal function and the renal biopsy findings.

DETAILED DESCRIPTION:
Using a prospective, randomised, open-labelled design, MP pulse treatment and cyclosporine A treatment will be compared for their efficacy in the treatment of severe HSP glomerulonephritis.

The trial will be a national multi-centre trial that involves all Finnish university hospitals, a few Finnish central hospitals.

The HSP patients with crescent HSP glomerulonephritis (ISKDC class III or IV) diagnosed by renal biopsy or with a renal biopsy finding of ISKDC class II + a distinct nephrotic syndrome will be included. Most of the patients will be recruited from a series collected by the same authors to study the prevention of HSP nephritis (see Effect of prednisone treatment on the symptoms of HSP disease and the development of glomerulonephritis).

The patients will be randomised to receive either MP pulses i.v. or cyclosporine A p.o. The MP pulses will consist of three doses of methylprednisolone 30 mg/kg i.v. given over a period of one week in hospital. On the intermediate days and for a month after the MP pulses, the patients will be given prednisone 30 mg/m2/day p.o., after which the prednisone medication will be gradually tapered over 3 months. The patients randomised into the cyclosporine A group will receive an initial dose of 5 mg/kg/day, after which the dosage will be titrated to an optimal therapeutic level by monitoring the B-Cya concentration. The cyclosporine A treatment will be continued for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* On the basis of a renal biopsy, the patient has been diagnosed for crescentic HSP glomerulonephritis of ISKDC grade III or IV or HSP glomerulonephritis of ISKDC grade II + a definite nephrotic syndrome (proteinuria > 40 mg/m2/h).

Exclusion Criteria:

* The child is on regular medication known to interact with cyclosporine. Such medication includes cisapride, phenytoin, phenobarbital, carbamazepine, digoxin and anti-inflammatory pain medication.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2000-01; Primary Completion 2007-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Disappearance of proteinuria/ hematuria | 24 mo
Renal function (measured by Cr-EDTA-Cl- GFR) | 24 mo
Renal biopsy findings | 24 mo

SECONDARY OUTCOMES:
Need for additional medication | 24 mo

CONTACTS AND LOCATIONS:
Overall Officials: Matti Nuutinen, M.D., Ph.D., Principal Investigator — Dept. of Pediatrics, Oulu University Hospital
Locations (1):
- Dept. of Pediatrics, Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Result] Jauhola O, Ronkainen J, Autio-Harmainen H, Koskimies O, Ala-Houhala M, Arikoski P, Holtta T, Jahnukainen T, Rajantie J, Ormala T, Nuutinen M. Cyclosporine A vs. methylprednisolone for Henoch-Schonlein nephritis: a randomized trial. Pediatr Nephrol. 2011 Dec;26(12):2159-66. doi: 10.1007/s00467-011-1919-5. Epub 2011 May 28. PMID 21626222
- [Derived] Hahn D, Hodson EM, Craig JC. Interventions for preventing and treating kidney disease in IgA vasculitis. Cochrane Database Syst Rev. 2023 Feb 28;2(2):CD005128. doi: 10.1002/14651858.CD005128.pub4. PMID 36853224